CLINICAL TRIAL: NCT04831372
Title: Comparing On-Table vs Off-Table Total Hip Arthroplasty Via the Direct Anterior Approach: A Prospective Randomized Trial
Brief Title: On-Table Versus Off-Table Total Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-1004
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Hip; Osteoarthritis, Hip
Keywords: Direct anterior approach; Hip arthroplasty; On table; Off table
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Primary Objectives- Determine whether there is a difference in operating room efficiency when preparing for, positioning, performing and turning over an operating room after a total hip arthroplasty (THA) via the direct anterior approach (DAA) when using a purpose built traction table ("On-Table") vs a standard operating table ("Off-Table")?
  Secondary Objective- Examine whether there is a difference in early post-operative pain, mobilization, complication rates and clinical outcomes when comparing patients who underwent a THA via the DAA when using an "On-Table" vs "Off-Table" technique.
Masking Description: BLINDING: none It is impossible to blind the surgeon to the arm as the techniques and instruments required for on-table vs off-table are substantially different. All subjects will be patients of Dr. Owen and he is the only operating surgeon for this study.
  The patient will see the beds when they are rolled into the operating room and are positioned. Thorough informed consent will make it apparent which table they are using.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On Table Group (Active Comparator): The Direct Anterior Approach (DAA) is a common way to perform total hip arthroplasty. There are two main techniques to perform total hip replacement through the anterior approach.
  The control group will be using the first method, which is the "on-table" method, which uses a specialized surgical table, called a traction table. This table involves placing both feet in specialized boots that are then hooked up to the table, and allows for positioning of the operative leg with aid of the table.
  Both the "on-table" and "off-table" techniques are routinely used both worldwide and by our joint replacement specialists at Carilion Clinic. This study will aim to compare the efficiency and efficacy of performing the DAA for total hip arthroplasty utilizing either the "on-table" or "off- table" technique. Patients will be randomized to receive their total hip arthroplasty with either the "on- table" or "off-table" method.
  Interventions: Procedure: On Table Group
- Off Table Group (Experimental): The Direct Anterior Approach (DAA) is a common way to perform total hip arthroplasty. There are two main techniques to perform total hip replacement through the anterior approach.
  The experimental group will be using the second method, which is the "off-table" method. In this method the patient is placed on a standard operating room table and the operative leg is manually positioned by the surgeon during the procedure . This obviates the need for the additional staff members or purchase of a specialized table.
  Both the "on-table" and "off-table" techniques are routinely used both worldwide and by our joint replacement specialists at Carilion Clinic. This study will aim to compare the efficiency and efficacy of performing the DAA for total hip arthroplasty utilizing either the "on-table" or "off- table" technique. Patients will be randomized to receive their total hip arthroplasty with either the "on- table" or "off-table" method.
  Interventions: Procedure: Off Table Group

INTERVENTIONS:
Procedure: Off Table Group — Total Hip arthroplasty being performed via the Direct Anterior Approach using a standard operating room table
  Arms: Off Table Group
Procedure: On Table Group — Total Hip arthroplasty being performed via the Direct Anterior Approach using a traction table
  Arms: On Table Group

SUMMARY:
The Direct Anterior Approach (DAA) is a common way to perform total hip arthroplasty. There are two main techniques to perform total hip replacement through the anterior approach. The first method is the "on-table" method, which uses a specialized surgical table, called a traction table. This table involves placing both feet in specialized boots that are then hooked up to the table, and allows for positioning of the operative leg with aid of the table. The major limitations associated with the traction table are the need for two additional staff members and the purchase of said table. The second method is the "off-table" method. In this method the patient is placed on a standard operating room table and the operative leg is manually positioned by the surgeon during the procedure . This obviates the need for the additional staff members or purchase of a specialized table. Both the "on-table" and "off-table" techniques are routinely used both worldwide and by our joint replacement specialists at Carilion Clinic. This study will aim to compare the efficiency and efficacy of performing the DAA for total hip arthroplasty utilizing either the "on-table" or "off- table" technique. Patients will be randomized to receive their total hip arthroplasty with either the "on- table" or "off-table" method.

DETAILED DESCRIPTION:
BACKGROUND: The Direct Anterior Approach (DAA) for total hip arthroplasty (THA) has become increasingly popular in the US over the last decade (Berry & Bozic, 2010). Major limitations of the DAA with traction table include the need for an additional surgeon's assistant, a traction table operator, and the purchase of said table. To counter these limitations, some surgeons advocate for the performing the DAA with a conventional operating room table {Cohen, 2017;Molenaers, 2017}. However to date, there are no studies directly comparing the efficiency and efficacy of these two techniques for DAA.

OBJECTIVE: Currently, it is unclear which surgical technique is more efficient and effective for total hip arthroplasties (THA). We hypothesize that there will be an increase in efficiency as measured by time when performing a standard operating table (Off-Table) DAA THA when compared to a purpose built traction table (On-Table) DAA THA. In addition, there will be less pain and faster functional recovery in the early post-operative period for patients who underwent an "Off-Table" DAA THA when compared to an "On-Table" DAA THA.

SPECIFIC AIMS: 1) Determine whether there is a difference in operating room efficiency between surgeries after a THA via DAA with a standard OR table versus a purpose-built traction table; 2) examine whether there is a difference in early post-operative pain and clinical outcomes when comparing patients who underwent a THA via the DAA with a standard OR table versus a purpose built traction table. 3) report differences in complication rates between those two.

METHODS: This is a prospective randomized clinical trial that will evaluate adult patients admitted to Carilion Clinic undergoing primary unilateral total hip arthroplasty. Off and on table DAA procedures will be performed by a single surgeon with multiple years of training and experience in both. Cluster randomization will be performed where patients will be randomized through scheduling. Demographic data will be collected. Operative records will be used to record operative times for each approach. Radiographs to assess implant positioning on postoperative day 0. The primary outcome variables are intra-operative data such as time the patient enters the operating room, time of incision, time of dressing application, exit room time, implants used, operative report. For secondary outcome variables, we will assess at 2 and 6 week follow ups routine Patient-Reported Outcome Measures including narcotic utilization based on pill count and MEq, and the PROMIS and HOOS, JR. measures.

EXPECTED OUTCOMES: We expect that the Off-table DAA technique will be associated with faster set up, surgical time, and overall room time when compared to the On-table approach. Additionally, we expect less early post-operative pain in the groin, knee and ankle. We expect that the patient report outcome measures at 2 and 6 weeks post-op for the off-table DAA group will be equivalent or better than the on-table DAA group. Finally we expect no difference in complication rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary unilateral THA
* Patient 18 years of age and older
* Patients who are able to provide consent

Exclusion Criteria:

* Bilateral procedure
* Non-Primary arthroplasty
* Prior non-arthroplasty operation requiring removal of hardware
* Inability to have spinal anesthesia (blood thinners)
* BMI > 40
* Active Smoking
* HbA1c > 8.0
* Failure to meet medical clearance
* Pregnant women per standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
Set Up Time | Time point that patient enters room to time point of first incision
  Time point that patient enters room to time point of first incision
Surgery Time | Time point of first incision to time point of dress application
  Time point of first incision to time point of dress application
Takedown Time | Time point of Dress application to Time point of exiting operating room
  Time point of Dress application to Time point of exiting operating room
Total Room Time | Time point that patient enters room to time point of exiting operating room
  Time point that patient enters room to time point of exiting operating room

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System/Hip Disability and Osteoarthritis Outcome Score, Joint Replacement scores | pre-op, 2 weeks post-op, 6 weeks post op, 1 year post op
  Hip pain measure survey on a scale of 0 - 10 with 0 = no pain and 10 = extreme pain
Visual Analog Scale scores | pre-op, 2 weeks post-op, 6 weeks post op, 1 year post op
  Hip, knee, ankle pain measure survey on a scale of 0 - 10 with 0 = no pain and 10 = worst pain
Narcotic Utillization | 2 weeks post op pill count
  Measured by pill count usage and converted into MME

CONTACTS AND LOCATIONS:
Overall Officials: Trevor M Owen, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Institute for Orthopaedics & Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to do so.

REFERENCES:
- [Background] Abdel MP, Berry DJ. Current Practice Trends in Primary Hip and Knee Arthroplasties Among Members of the American Association of Hip and Knee Surgeons: A Long-Term Update. J Arthroplasty. 2019 Jul;34(7S):S24-S27. doi: 10.1016/j.arth.2019.02.006. Epub 2019 Feb 12. PMID 30852068
- [Background] Bender B, Nogler M, Hozack WJ. Direct anterior approach for total hip arthroplasty. Orthop Clin North Am. 2009 Jul;40(3):321-8. doi: 10.1016/j.ocl.2009.01.003. PMID 19576399
- [Background] Berger RA. Mini-incision total hip replacement using an anterolateral approach: technique and results. Orthop Clin North Am. 2004 Apr;35(2):143-51. doi: 10.1016/S0030-5898(03)00111-1. PMID 15062700
- [Background] Berry DJ, Bozic KJ. Current practice patterns in primary hip and knee arthroplasty among members of the American Association of Hip and Knee Surgeons. J Arthroplasty. 2010 Sep;25(6 Suppl):2-4. doi: 10.1016/j.arth.2010.04.033. Epub 2010 Jul 1. PMID 20580196
- [Background] Cohen EM, Vaughn JJ, Ritterman SA, Eisenson DL, Rubin LE. Intraoperative Femur Fracture Risk During Primary Direct Anterior Approach Cementless Total Hip Arthroplasty With and Without a Fracture Table. J Arthroplasty. 2017 Sep;32(9):2847-2851. doi: 10.1016/j.arth.2017.04.020. Epub 2017 Apr 21. PMID 28511947
- [Background] Matta JM, Shahrdar C, Ferguson T. Single-incision anterior approach for total hip arthroplasty on an orthopaedic table. Clin Orthop Relat Res. 2005 Dec;441:115-24. doi: 10.1097/01.blo.0000194309.70518.cb. PMID 16330993
- [Background] Molenaers B, Driesen R, Molenaers G, Corten K. The Direct Anterior Approach for Complex Primary Total Hip Arthroplasty: The Extensile Acetabular Approach on a Regular Operating Room Table. J Arthroplasty. 2017 May;32(5):1553-1559. doi: 10.1016/j.arth.2016.12.016. Epub 2016 Dec 22. PMID 28087159
- [Background] Nakata K, Nishikawa M, Yamamoto K, Hirota S, Yoshikawa H. A clinical comparative study of the direct anterior with mini-posterior approach: two consecutive series. J Arthroplasty. 2009 Aug;24(5):698-704. doi: 10.1016/j.arth.2008.04.012. Epub 2008 Jun 13. PMID 18555653
- [Background] Post ZD, Orozco F, Diaz-Ledezma C, Hozack WJ, Ong A. Direct anterior approach for total hip arthroplasty: indications, technique, and results. J Am Acad Orthop Surg. 2014 Sep;22(9):595-603. doi: 10.5435/JAAOS-22-09-595. PMID 25157041
- [Background] Restrepo C, Parvizi J, Pour AE, Hozack WJ. Prospective randomized study of two surgical approaches for total hip arthroplasty. J Arthroplasty. 2010 Aug;25(5):671-9.e1. doi: 10.1016/j.arth.2010.02.002. Epub 2010 Apr 8. PMID 20378307
- [Background] Tian S, Goswami K, Manrique J, Blevins K, Azboy I, Hozack WJ. Direct Anterior Approach Total Hip Arthroplasty Using a Morphometrically Optimized Femoral Stem, a Conventional Operating Table, Without Fluoroscopy. J Arthroplasty. 2019 Feb;34(2):327-332. doi: 10.1016/j.arth.2018.10.023. Epub 2018 Oct 26. PMID 30448326